## NCT03464422

Title of Research Project: Adapting an Evidence-based Intervention for Stigma-related Stress, Mental Health, and HIV Risk for MSM of Color in Small Urban Areas (ESTEEM-conneCT)

SAP Date 6.3.2021

## Adapting an Evidence-based Intervention for Stigma-related Stress, Mental Health, and HIV Risk for MSM of Color in Small Urban Areas (ESTEEM-conneCT)

## Statistical Analysis Plan

After computing descriptive statistics of demographic and outcome variables, we performed t-tests to assess changes in stigma-related stress—to capture any improvements in stigma coping—comparing mean baseline scores with mean 3-month post-treatment scores. We similarly examined pre-post changes in mental and sexual health. We focus our quantitative analysis on effect sizes and an examination of the overall pattern of changes, as this pilot investigation is not powered to detect significant treatment effects, does not rely on a clinical sample, and is not intended to serve as a test of treatment efficacy. We calculated Hedge's g effect sizes to highlight the relative effect sizes across study outcomes because, unlike Cohen's d, Hedge's g provides unbiased estimates, even for smaller samples (n < 20; Lakens, 2013).

## References

Lakens, D. (2013). Calculating and reporting effect sizes to facilitate cumulative science: a practical primer for t-tests and ANOVAs. Frontiers in psychology, 4, 863.